CLINICAL TRIAL: NCT00171977
Title: Post-Marketing Clinical Study of Postoperative Adjuvant Therapy With Imatinib Mesylate in Patients With Gastrointestinal Stromal Tumors (GIST)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSTI571BJP07
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2012-08-07 (Estimated); Status verified 2012-08

CONDITIONS: Gastrointestinal Stromal Tumors
Keywords: GIST; Imatinib; Postoperative Adjuvant
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — Imatinib Mesylate

ARMS (1):
- Imatinib Mesylate (Experimental): 400 mg once per day
  Interventions: Drug: Imatinib Mesylate

INTERVENTIONS:
Drug: Imatinib Mesylate
  Other Names: Gleevec/Glivec; STI571

SUMMARY:
This is a multicenter, post-marketing, clinical study evaluating the safety and efficacy of postoperative adjuvant therapy with Imatinib Mesylate in high-risk patients after curative resection of newly diagnosed GIST.Patients will be evaluated for relapse -free survival as measured by the confirmation of tumor recurrence and survival for 3 years after surgery for their primary tumors.

ELIGIBILITY:
Inclusion Criteria:

* underwent macroscopically curative resection;
* immunohistochemically confirmed KIT (CD117)-positive tumors;
* judged as being high-risk according to the criteria for risk classification

Exclusion Criteria:

* synchronous double cancer or metachronous double cancer with a disease-free period of ≤5 years;
* received therapy with Imatinib Mesylate prior to study entry;
* cardiac problem of Grade 3 or higher (New York Heart Association (NYHA) criteria)

Other protocol-defined inclusion / exclusion criteria may apply.

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2004-07; Primary Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
To evaluate the relapse-free survival (RFS) in patients receiving postoperative adjuvant therapy | 3 years

SECONDARY OUTCOMES:
To evaluate overall survival, relapse free | 3 years
Safety | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Tokyo, Japan

REFERENCES:
- [Derived] Kanda T, Nishida T, Wada N, Kobayashi O, Yamamoto M, Sawaki A, Boku N, Koseki M, Doi T, Toh Y, Kakeji Y, Sugiyama T, Komatsu Y, Kikuchi S, Ogoshi K, Katai H, Miyachi K, Hirota S, Ohtsu A. Adjuvant therapy with imatinib mesylate after resection of primary high-risk gastrointestinal stromal tumors in Japanese patients. Int J Clin Oncol. 2013 Feb;18(1):38-45. doi: 10.1007/s10147-011-0339-7. Epub 2011 Nov 23. PMID 22105894
- [Derived] Essat M, Cooper K. Imatinib as adjuvant therapy for gastrointestinal stromal tumors: a systematic review. Int J Cancer. 2011 May 1;128(9):2202-14. doi: 10.1002/ijc.25827. PMID 21387287